CLINICAL TRIAL: NCT01611493
Title: A Prospective, Randomized-Controlled Evaluation of the Osseotite CP4 Certain Prevail Tapered Implant for the Preservation of Crestal Bone
Brief Title: Osseotite Certain Prevail for the Preservation of Crestal Bone
Acronym: OCPTI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andres Duque Duque (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor-Investigator, Andres Duque Duque, Principal investigator, CES University
Organization: CES University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: implantes3i
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Dental Implants; Jaw, Edentulous, Partially/rehabilitation; Jaw, Edentulous, Partially/surgery; randomised Clinical Trials; Humans
MeSH Terms: conditions — Jaw, Edentulous, Partially; Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osseotite Prevail Implant (Experimental): The Osseotite Prevail will be placed in sites with native bone, with at least three months of healing since tooth extraction or four months from bone augmentation grafting procedure.
  Interventions: Device: Osseotite Prevail Implant
- Osseotite Non Prevail Implant (Active Comparator): Osseotite Non Prevail Implant will be placed in sites with native bone, with at least three months of healing since tooth extraction or four months from bone augmentation grafting procedure
  Interventions: Device: Osseotite Non Prevail Implant

INTERVENTIONS:
Device: Osseotite Prevail Implant — Osseotite Prevail will be placed in sites with native bone, with at least three months of healing since tooth extraction or four months from bone augmentation grafting procedure
  Arms: Osseotite Prevail Implant
Device: Osseotite Non Prevail Implant — Osseotite Non Prevail Implant will be placed in sites with native bone, with at least three months of healing since tooth extraction or four months from bone augmentation grafting procedure
  Arms: Osseotite Non Prevail Implant

SUMMARY:
A potential complicating factor affecting implants is crestal bone loss. The causes of crestal bone loss are attributed to several factors. Among those hypothesized, proof for one or another cause remains obscure. Clinical documentation suggests that implant design may be a key factor. While the evidence is inconclusive, various authors suggest that it is a result of a combination of effects including (1) limited drilling procedure and restricted second-stage surgery 2, (2) rough implant surface in crestal bone 3, (3) microthread design for implant stiffness 4, (4) loading along a conus versus a flat interface 5, and (5) the absence of a significant microgap 6.

The practice of platform switching (e.g. placing a 4 mm diameter abutment on a 5 mm implant seating surface physically moves the inflammatory cell infiltrate zone away from the crestal bone). The growing body of anecdotal platform switch evidence supports this biological width hypothesis. Here the biological width refers to the height of the dento-gingival attachment apparatus around a normal tooth and is defined as the distance necessary for a healthy existence of bone and soft tissue from the most apical extent of a dental restoration.

To formally test this hypothesis the current study has been designed. The Prevail implant has been made with an integrated medialized seating surface that establishes a platform switching function. This implant moves the implant/abutment interface away from the crestal bone and may therefore reduce the amount of bone loss observed in the standard (non-medialized) Osseotite implant design. The objective of this study is to evaluate crestal bone levels adjacent to the implant reference point from the time of implant placement to a period of two years after loading.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex and any race greater than 18 years of age
* Patients for whom a decision has already been made to use dental implants for the restoration of existing edentulism in the mandible or maxilla.
* Patients must be physically able to tolerate conventional surgical and restorative procedures.
* Patients must agree to be evaluated for each study visit, especially the yearly follow-up visits.

Exclusion Criteria:

* Patients with active infection or severe inflammation in the areas intended for implant placement.
* Patients with a > 10 cigarette per day smoking habit.
* Patients with uncontrolled diabetes mellitus.
* Patients with uncontrolled metabolic bone disease where there is a diagnosis of the following: Osteomalacia, primary or secondary hyperparathyroidism, renal osteodystrophy, or Paget's disease of bone.
* Patients with a history of therapeutic radiation to the head
* Patients in need of bone grafting at the site of the intended study implant for augmentation purposes.
* Patients who are known to be pregnant at the screening visit.
* Patients with evidence of severe para-functional habits such as bruxing or clenching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-11 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Preservation of crestal bone | Two years

SECONDARY OUTCOMES:
Osseus integration | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Andres Duque, MSc, Principal Investigator — CES University; Pablo E Correa, MSc, Principal Investigator — CES University; Astrid Giraldo, Postgraduate, Principal Investigator — CES University
Locations (1):
- CES University / Faculty of Dentistry, Medellín, Antioquia, Colombia